CLINICAL TRIAL: NCT02786160
Title: The Effects of Human Milk Oligosaccharides (HMO) on the Faecal Microbiota and on Host Metabolism in Obese Children: A Parallel, Double-blind, Randomized, Placebo-controlled Study
Brief Title: Effects of HMOs on the Faecal Microbiota and on Host Metabolism in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycom A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NATROB; SJ-528 (Other: Den Videnskabsetiske Komité for Region Sjaelland)
Record Dates: First submitted 2016-05-23; First posted 2016-05-30 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Health Maintenance Organizations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HMO1 (Active Comparator): Daily bolus of HMO1
  Interventions: Dietary Supplement: HMO
- HMO2 (Active Comparator): Daily bolus of HMO2
  Interventions: Dietary Supplement: HMO
- Dextropur (Placebo Comparator): Daily bolus of Dextropur
  Interventions: Dietary Supplement: Dextropur

INTERVENTIONS:
Dietary Supplement: HMO
  Arms: HMO1; HMO2
Dietary Supplement: Dextropur
  Arms: Dextropur

SUMMARY:
The study is a randomised, placebo-controlled, double-blind, parallel study in obese children. A total of 75 obese children in the age 5 to 10 years, enrolled in a childhood obesity treatment program, will be included. The participating children will be randomised into one of three groups consuming either HMO (two groups) or placebo (one group).

The primary objective of the study is to establish the effects of HMOs on the faecal microbiota in children. Secondary objectives are to evaluate safety of HMO supplementation in children and the effect on gastrointestinal symptoms (tolerance), bowel habits, metabolic profile and body composition in obese children.

ELIGIBILITY:
Inclusion Criteria:

1. Informed, written consent by the child's representative(s) and informed verbal assent by the child
2. Age ≥5 and <11 years at visit 0
3. BMI SDS of ≥ 2.3
4. Enrolment in the childhood obesity treatment program at the Children's Obesity Clinic
5. Ability and willingness to understand and comply with the study procedures
6. The child's representative(s) need(s) to read, speak and understand Danish

Exclusion Criteria:

1. Participation in another clinical intervention study one month prior to the screening visit and throughout the study.
2. Any gastrointestinal disease(s) that may cause symptoms or may interfere with the trial outcome, as judged by the investigator.
3. Other severe disease(s) such as malignancy, kidney disease or neurological disease, as judged by the investigator.
4. Psychiatric disease, as judged by the investigator.
5. Use of probiotic supplements (yoghurt allowed) 3 months prior to screening and throughout the study.
6. Consumption of antibiotic drugs 3 months prior to screening and throughout the study.
7. Consumption on a regular basis of medication that might interfere with symptom evaluation (as judged by the investigator) 2 weeks prior to screening and throughout the study.
8. Lack of suitability for participation in the study for any reason as judged by the investigator.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in faecal microbiota profile | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out

SECONDARY OUTCOMES:
Change from baseline in clinical chemistry | Baseline and after 8 weeks of intake, and after 10 months of wash-out
Change from baseline in haematology | Baseline and after 8 weeks of intake, and after 10 months of wash-out
Change from baseline in gastrointestinal symptoms measured via the gastrointestinal symptom rating scale (GSRS) | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out
Change from baseline in Bristol Stool Form Scale (BSFS) | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out
Change from baseline in specific host-bacteria metabolic biomarkers in blood | Baseline and after 8 weeks of intake, and after 10 months of wash-out
Change from baseline of HOMA-IR | Baseline and after 8 weeks of intake, and after 10 months of wash-out
Change from baseline of BMI-SDS | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out
Change from baseline of fat percentage | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out
Change from baseline of waist circumference | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out
Change from baseline of hip circumference | Baseline and after 4 and 8 weeks of intake, and after 2 and 10 months of wash-out
Change from baseline of specific blood biomarkers related to gut barrier function | Baseline and after 8 weeks of intake, and after 10 months of wash-out
Change from baseline of specific blood biomarkers related to inflammation | Baseline and after 8 weeks of intake, and after 10 months of wash-out
Change from baseline of specific faecal biomarkers related to inflammation | Baseline and after 8 weeks of intake, and after 10 months of wash-out

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Christian Holm, MD, PhD, Principal Investigator — Holbaek Hospital
Locations (1):
- Department of Paediatrics, Holbaek Hospital, Holbæk, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fonvig CE, Amundsen ID, Vigsnaes LK, Sorensen N, Frithioff-Bojsoe C, Christiansen M, Hedley PL, Holm LA, McConnell B, Holm JC. Human Milk Oligosaccharides Modulate Fecal Microbiota and Are Safe for Use in Children With Overweight: A Randomized Controlled Trial. J Pediatr Gastroenterol Nutr. 2021 Sep 1;73(3):408-414. doi: 10.1097/MPG.0000000000003205. PMID 34139746